CLINICAL TRIAL: NCT02482961
Title: Prospective Observational Study, Impact of Plasma Levels of Colistin in Patients With Carbapenem Resistant Acinetobacter Baumannii Infection
Brief Title: Impact of Plasma Levels of Colistin in Patients With Carbapenem Resistant Acinetobacter Baumannii Infection
Status: Completed | Type: Observational
Sponsor: DongGuk University (Other)
Responsible Party: Principal Investigator, Young Soon Yoon, assistant professor, DongGuk University
Other Study IDs: 2014-128
Record Dates: First submitted 2015-06-03; First posted 2015-06-26 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Acinetobacter Infections
MeSH Terms: conditions — Acinetobacter Infections | interventions — colistinmethanesulfonic acid; Colistin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: colistimethate sodium — At least once a week, all patients with carbapenem-resistant Acinetobacter baumannii infection were screened from the database at the clinical microbiology laboratory
  Other Names: colistin

SUMMARY:
This study purposed to examine the adequate range of therapeutic concentration for Korean people by observing curative effects, side effects, blood concentration, etc. in treating CRAB-infected patients with colistin.

DETAILED DESCRIPTION:
Acinetobacter baumanii usually causes pneumonia and sepsis, and is susceptible to antibiotics such as ampicillin/sulbactam and carbapenem, but it easily becomes tolerant and there are few other drugs usable. Particularly in Korean patients with ventilator-associated pneumonia (VAP), the percentage of carbapenem-resistant Acinetobacter baumannii (CRAB) is increasing recently.

Colistin (polymyxin E) is antibiotic of polymyxin line used to multidrug-resistant gram-negative bacteria such as Klebsiella pneumonia, Pseudomonas aeruginosa, and Acinetobacter baumannii, and it produces bactericidal action by destroying bacterial cell membrane. Colistin was antibiotic isolated from Bacillius polymyxa subspecies colistinus first in Japan in 1949, and has long been used in clinic since 1959, but its use through intravenous infusion decreased in the 1970s due to acute kidney injury and neurotoxicity. Recently, however, it is being used more frequently for hospital infection by multidrug-resistant gram-negative bacteria and, as a result, various studies are being conducted on colistin.

Colistin consists of over 30 different polymyxin compounds including colistin A (polymyxin E1) and colistin B (polymyxin E2), and colistimethate sodium (CMS) and colistin sulfate are used. In Korea, it is usually administered intravenously in the form of CMS, which is an inactive precursor. In the body, CMS is metabolized into various metabolites including colistin or is discharged through urine. In contrast, active metabolite colistin is hardly discharged through urine, and is removed through non-renal elimination, but the accurate extracorporeal elimination mechanism is still unknown. CMS reaches the peak serum concentration in 10 minutes from intravenous administration, and its half-life is 2.2 hours while the half-life of colistin 18.5 hours.

With regard to the bactericidal activity of colistin, the unbound area under the concentration-time curve/minimum inhibitory concentration (fAUC/MIC) is important, and adequate exposure to the drug has been known to be important for curative effect, but it is still controversial what the optimal dose and interval are. Although the drug has been used long, the accurate measuring of colistin blood concentration became possible only in the mid 2000s and, therefore, pharmacokinetic research on the drug has been conducted relatively recently and there is increasing interest in the validity of established uses, adequate uses, therapeutic drug monitoring, etc. Two of the established uses of the drug are intravenous administration of 2.5~5mg/kg/day divided into 2~4 times to patients with normal renal function, adjusting the dose and interval of administration according to renal function (package insert), and the administration of loading dose followed by 2~3 times of administration depending on renal function. The major side effects of colistin are nephrotoxicity and neurotoxicity, and according to a recent study, the incidence of nephrotoxicity caused by colistin was 30~60%. Renal insufficiency is more frequent when vancomycin is used together in VAP. Renal insufficiency is known to be reversible, but some cases require dialysis. Known risk factors of renal insufficiency include cumulative CMS dose, combined use of drugs inducing renal insufficiency, female, and age.

There have been ex vivo studies for assessing the bactericidal effect of colistin for exploring its adequate uses and case studies for evaluating the risk factors of nephrotoxicity, one of the major side effects yet there are still controversial issues related to the drug. Furthermore, as most of these studies were conducted with Western subjects, their results are hardly applicable to Koreans as they are. Thus, this study purposed to examine the adequate range of therapeutic concentration for Korean people.

ELIGIBILITY:
Inclusion Criteria:

1. All adult patients (aged ≥18 years)
2. Microbiological evidence (sputum, urine, blood) of infection due to carbapenem-resistant Acinetobacter baumannii during hospitalization
3. Intravenous Colistimethate sodium treated patient with Acinetobacter baumannii infection who fulfill the above criteria
4. Patients who agree to the gathering clinical information by means of an informed consent

Exclusion Criteria:

1. Pregnancy and lactating women
2. Patients receiving Colistimethate sodium therapy for <48 hours
3. Patient of chronic renal disease defined as a Creatinine clearance <10 mL/min, Or requirement for peritoneal or hemo-dialysis or hemofiltration
4. Known hypersensitivity to Colistimethate sodium
5. Receiving intravenous colistin therapy within the past 30 days
6. Patients treated with nebulized Colistimethate sodium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients (aged ≥18 years)had Microbiological evidence (sputum, urine, blood) of infection due to carbapenem-resistant Acinetobacter baumannii result during the study period at Dongguk University Ilsan Hospital
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-05; Primary Completion 2018-01-10 (Actual); Study Completion 2018-04-04 (Actual)

PRIMARY OUTCOMES:
Difference in plasma drug concentration between patients with nephrotoxicity and those without | Participants will be followed for the duration of hospital stay, an expected average of 2-3wks. Nephrothoxicity was determined during colistin use.
  - Criteria for diagnosing nephrotoxicity: Creatinine clearance (CrCL) decreases to 50% of the baseline value or serum creatinine concentration (SCr) doubles, or renal replacement therapy is required.

SECONDARY OUTCOMES:
Difference in plasma drug concentration between patients showing clinical cure or improvement and those of treatment failure | Participants will be followed for the duration of hospital stay, an expected average of 2-3wks. Clinical outcome was determined at the final day of colistin use.
  Criteria for clinical cure/improvement:
  * Clinical cure: The symptoms and signs of infection have disappeared completely at the end of treatment.
  * Clinical improvement: The symptoms and signs of infection have disappeared partially at the end of treatment.
Difference in plasma drug concentration according to microbiological response | Participants will be followed for the duration of hospital stay, an expected average of 2-3wks.
  - Microbiological response: Pathogens are not cultured at the end of treatment.
Difference in plasma drug concentration according to in-hospital mortality | Participants will be followed for the duration of hospital stay, an expected average of 2-5wks.
Difference in plasma drug concentration according to the RIFLE Criteria for nephrotoxicity | Participants will be followed for the duration of hospital stay, an expected average of 2-3wks.
Risk factors associated with nephrotoxicity | Participants will be followed for the duration of hospital stay, an expected average of 2-3wks.
  Use of NSAIDS or other antibiotics, age and sex etc. associated with nephrotoxicity will be analyzed.
Difference in plasma drug concentration between patients with abnormality of liver function. | Participants will be followed for the duration of hospital stay, an expected average of 2-3ks.
Difference in plasma drug concentration between patients with abnormality of thrombocytopenia. | Participants will be followed for the duration of hospital stay, an expected average of 2-3ks.
Difference in plasma drug concentration between patients with abnormality of neuropathy. | Participants will be followed for the duration of hospital stay, an expected average of 2-3ks.

CONTACTS AND LOCATIONS:
Overall Officials: Young-Soon Yoon, professor, Study Chair — DongGuk University
Locations (1):
- Dongguk University Ilsan Hospital, Goyang, Kyonggido, South Korea

REFERENCES:
- [Derived] Jeong YJ, Gu N, Kwack WG, Kang Y, Park SY, Yoon YS. Prospective observational study of the impact of plasma colistin levels in patients with carbapenem-resistant Acinetobacter baumannii pneumonia. J Glob Antimicrob Resist. 2021 Dec;27:315-323. doi: 10.1016/j.jgar.2021.10.017. Epub 2021 Nov 12. PMID 34775134